CLINICAL TRIAL: NCT01542190
Title: A Randomized, Masked Comparison of Topical Ketorolac 0,4% Versus Placebo in Cataract Surgery.
Brief Title: Comparison of Topical Ketorolac 0,4% Versus Placebo in Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Joao Paulo Felix, Dr., University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0018014600011
Record Dates: First submitted 2012-02-07; First posted 2012-03-02 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Cystoid Macular Edema Following Cataract Surgery, Bilateral
Keywords: cataract surgery; cystoid macular edema; angiography
MeSH Terms: conditions — Macular Edema | interventions — Ketorolac Tromethamine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ketorolac tromethamine (Active Comparator)
  Interventions: Drug: Ketorolac Tromethamine
- Dextrano 70 / Hypromellose (Placebo Comparator)
  Interventions: Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Ketorolac Tromethamine — ketorolac tromethamine 0.4%
  Other Names: Acular LS (Allergan); Lacribell (Latinofarma)

SUMMARY:
The purpose of this study is to compare effects of preoperative and postoperative use of topical ketorolac tromethamine 0.4% versus placebo in uncomplicated cataract surgery.

Patients scheduled to undergo phacoemulsification will be randomized to receive either topical prednisolone acetate 1% 4 times daily (QID) plus dextran 70/hypromellose QID (placebo group) or topical prednisolone 1% QID plus ketorolac tromethamine 0.4% QID (ketorolac group) for three days preoperatively and four weeks postoperatively. The primary outcome 5 weeks after surgery will be angiographic cystoid macular edema.

DETAILED DESCRIPTION:
Purpose:

To compare effects of preoperative and postoperative use of topical ketorolac tromethamine 0.4% versus placebo in uncomplicated cataract surgery.

Methods:

This will be a masked single-center, randomized clinical study comprising 80 patients undergoing phacoemulsification cataract surgery. Patients scheduled to undergo phacoemulsification and with no recognized cystoid macular edema (CME) risks (diabetic retinopathy, retinal vascular disease or macular abnormality) will be randomized to receive either topical prednisolone acetate 1% 4 times daily (QID) plus dextran 70/hypromellose QID (placebo group;n=40) or topical prednisolone 1% QID plus ketorolac tromethamine 0.4% QID (ketorolac group;n=40) for three days preoperatively and four weeks postoperatively. In both groups topical gatifloxacin will be administered to the treated eye QID, starting three days before surgery and continuing for seven days. The primary outcome 5 weeks after surgery will be angiographic cystoid macular edema. Other included outcomes will be best corrected visual acuity (BCVA), intraocular pressure (IOP), CME incidence, retinal thickness as measured by spectral-domain optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with nuclear cataract, density 1 and 2 classified by LOCS II, scheduled to undergo phacoemulsification cataract surgery.

Exclusion Criteria:

* Patients with:

  * Diabetes,
  * Hypertension,
  * uveitis,
  * macular disease,
  * congenital ocular abnormalities,
  * cataract density 0 and 3 by LOCS II,
  * pseudoexfoliation syndrome.

Patients under treatment with nonsteroidal antinflammatory drugs or topical eye drops were excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
cystoid macular edema | 1 month
  Angiography (Miyake's criteria)

SECONDARY OUTCOMES:
Best corrected visual acuity | 1 month
  ETDRS.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo PC Lira, Study Chair — University of Campinas, Brazil
Locations (1):
- Unicamp, Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Miyake K, Masuda K, Shirato S, Oshika T, Eguchi K, Hoshi H, Majima Y, Kimura W, Hayashi F. Comparison of diclofenac and fluorometholone in preventing cystoid macular edema after small incision cataract surgery: a multicentered prospective trial. Jpn J Ophthalmol. 2000 Jan-Feb;44(1):58-67. doi: 10.1016/s0021-5155(99)00176-8. PMID 10698027
- [Background] Miyake K, Ibaraki N. Prostaglandins and cystoid macular edema. Surv Ophthalmol. 2002 Aug;47 Suppl 1:S203-18. doi: 10.1016/s0039-6257(02)00294-1. PMID 12204717
- [Background] Kim A, Stark WJ. Are topical NSAIDs needed for routine cataract surgery? Am J Ophthalmol. 2008 Oct;146(4):483-5. doi: 10.1016/j.ajo.2008.07.027. No abstract available. PMID 18804560
- [Background] Gass JD, Norton EW. Cystoid macular edema and papilledema following cataract extraction. A fluorescein fundoscopic and angiographic study. Arch Ophthalmol. 1966 Nov;76(5):646-61. doi: 10.1001/archopht.1966.03850010648005. No abstract available. PMID 5955948
- [Background] Miyake K. Prevention of cystoid macular edema after lens extraction by topical indomethacin (I). A preliminary report. Albrecht Von Graefes Arch Klin Exp Ophthalmol. 1977 Aug 8;203(2):81-8. doi: 10.1007/BF00413399. PMID 303062
- [Background] Miyake K, Ota I, Miyake G, Numaga J. Nepafenac 0.1% versus fluorometholone 0.1% for preventing cystoid macular edema after cataract surgery. J Cataract Refract Surg. 2011 Sep;37(9):1581-8. doi: 10.1016/j.jcrs.2011.03.052. PMID 21855758
- [Background] Rossetti L, Chaudhuri J, Dickersin K. Medical prophylaxis and treatment of cystoid macular edema after cataract surgery. The results of a meta-analysis. Ophthalmology. 1998 Mar;105(3):397-405. doi: 10.1016/S0161-6420(98)93018-4. PMID 9499767
- [Background] Wittpenn JR, Silverstein S, Heier J, Kenyon KR, Hunkeler JD, Earl M; Acular LS for Cystoid Macular Edema (ACME) Study Group. A randomized, masked comparison of topical ketorolac 0.4% plus steroid vs steroid alone in low-risk cataract surgery patients. Am J Ophthalmol. 2008 Oct;146(4):554-560. doi: 10.1016/j.ajo.2008.04.036. Epub 2008 Jul 2. PMID 18599019
- See also: Estate University of Campinas — http://www.fcm.unicamp.br